CLINICAL TRIAL: NCT05659004
Title: The Experiences of Patients With Chronic Limb-threatening Ischaemia From First Symptom to Vascular Surgery Assessment: a Qualitative Study
Brief Title: Referrals for CLTI: Qualitative Study
Status: Completed | Type: Observational
Sponsor: University of Hull (Other)
Collaborators: The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Other Study IDs: 321794
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Limb Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: 1 qualitative interview
  Interventions: Behavioral: Qualitative interview

INTERVENTIONS:
Behavioral: Qualitative interview — No intervention

SUMMARY:
The goal of this qualitative study is to explore the experiences of patients who have been diagnosed with chronic limb-threatening ischaemia (CLTI). The main questions it aims to answer are:

* What are the perceptions and experiences of patients between first symptom of CLTI and vascular surgery assessment
* What is important to patients during this process.

Participants will be interviewed and their words analysed using reflexive thematic analysis.

DETAILED DESCRIPTION:
There are delays at every stage of the patient journey from developing chronic limb-threatening ischaemia (CLTI) to treatment, associated with poorer outcomes for patients. There is currently limited national and international guidance on how and when to refer patients with suspected CLTI to specialist vascular surgery services. The use of qualitative interviews will allow us explore perceptions and experiences of patients with CLTI being referred to vascular surgery services, and identify possible ways to improve the process via interviews. This study will provide novel information on patient experience, and together with other work provide a framework for improvement of the referral process for CLTI.

ELIGIBILITY:
Inclusion Criteria:

- CLTI diagnosed in the last year

Exclusion Criteria:

* Lacking capacity to consent to interview
* Potential to be violent
* Cognitive impairment
* Non-English speaking

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic limb-threatening ischaemia in the last year
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Experiences and perceptions of patients on their journey to diagnosis of CLTI | To be conducted in 2023
  Exploring patient experience

SECONDARY OUTCOMES:
Potential improvements the process from first symptom to diagnosis of CLTI | To be conducted in 2023
  Identifying targets for improvement work

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chetter, MD, Study Director — University of Hull
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Trust, Cambridge, Cambd
  - Mid Yorkshire Hospitals NHS Trust, Wakefield, Yorkshire

IPD SHARING:
Plan to Share IPD: No
There is no plan; data will not be shared.